CLINICAL TRIAL: NCT00676338
Title: Safety and Efficacy of Exenatide Once Weekly Injection Versus Metformin, Dipeptidyl Peptidase-4 Inhibitor, or Thiazolidinedione as Monotherapy in Drug-Naive Patients With Type 2 Diabetes
Brief Title: Safety and Efficacy of Exenatide Once Weekly Injection Versus Metformin, Dipeptidyl Peptidase-4 Inhibitor, or Thiazolidinedione as Monotherapy in Drug-Naive Patients With Type 2 Diabetes (DURATION-4)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H8O-MC-GWCH (DURATION - 4)
Record Dates: First submitted 2008-05-09; First posted 2008-05-13 (Estimated); Results first posted 2012-11-26 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2015-03

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Amylin; Lilly; exenatide once weekly; Byetta; Januvia; sitagliptin; thiazolidinedione
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin; Sitagliptin Phosphate; Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Exenatide Once Weekly (Experimental)
  Interventions: Drug: exenatide once weekly
- Metformin (Active Comparator)
  Interventions: Drug: metformin
- Sitagliptin (Active Comparator)
  Interventions: Drug: sitagliptin
- Pioglitazone (Active Comparator)
  Interventions: Drug: pioglitazone

INTERVENTIONS:
Drug: exenatide once weekly — subcutaneous injection, 2mg, once weekly plus placebo oral once daily
  Arms: Exenatide Once Weekly
Drug: metformin — oral, 1000-2500mg, daily plus placebo once weekly subcutaneous injection
  Arms: Metformin
Drug: sitagliptin — oral, 100 mg, daily plus placebo once weekly subcutaneous injection
  Arms: Sitagliptin
Drug: pioglitazone — oral, 30-45mg, daily plus placebo once weekly subcutaneous injection
  Arms: Pioglitazone

SUMMARY:
This study will compare the effects of 2.0 mg exenatide once weekly injection as monotherapy to 3 active comparators(metformin, dipeptidyl peptidase-4 inhibitor, and thiazolidinedione) in drug naive patients with type 2 diabetes treated with diet and exercise.

ELIGIBILITY:
Inclusion Criteria:

* have type 2 diabetes and are treated with diet and exercise alone.
* at least 18 years of age.
* HbA1c between 7.1% and 11.0%, inclusive.
* Body mass index (BMI) of 23 kg/m2 to 45 kg/m2, inclusive.
* Have a history of stable body weight (not varying by >5% for at least 3 months prior to screening).

Exclusion Criteria:

* Have history of cardiac disease or presence of active cardiac disease within the year prior to inclusion in the study including myocardial infarction, clinically significant arrhythmia, unstable angina, moderate to severe congestive heart failure, coronary artery bypass surgery, or angioplasty
* Have a history of renal transplantation or are currently receiving renal dialysis
* Have active or untreated malignancy, or have been in remission from clinically significant malignancy (other than basal cell or squamous cell skin cancer, in situ carcinomas of the cervix, or in situ prostate cancer) for less than 5 years.
* Have history of severe GI disorder (e.g., gastroparesis)
* Have a history of acute or chronic pancreatitis.
* Have active proliferative retinopathy.
* Have been treated with drugs that promote weight loss (e.g., Xenical®[orlistat], Meridia® [sibutramine], Acomplia® [rimonabant], Acutrim® [phenylpropanolamine], or similar over-the-counter medications) within 3 months of screening.
* Have been treated with any antidiabetic agent for more than 7 days within 3 months prior to screening.
* Have had an organ transplant.
* Have previously completed or discontinued study drug in this study, withdrawn from this study or any other study investigating exenatide once weekly.
* Have received treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry.
* Are currently enrolled in any other clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 820 (Actual)
Dates: Start 2008-11; Primary Completion 2010-07 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, MD, Study Director — Eli Lilly and Company
Locations (106):
- United States (18):
  - Research Site, Buena Park, California
  - Research Site, Los Angeles, California
  - Research Site, Valencia, California
  - Research Site, Jacksonville, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Meridian, Idaho
  - Research Site, Des Moines, Iowa
  - Research Site, Grand Rapids, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, Billings, Montana
  - Research Site, Toms River, New Jersey
  - Research Site, Wilmington, North Carolina
  - Research Site, Danville, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Wilke Barre, Pennsylvania
  - Research Site, Austin, Texas
  - Research Site, El Paso, Texas
  - Research Site, New Branufels, Texas
- Argentina (2):
  - Research Site, Buenos Aires
  - Research Site, Mar del Plata
- Belgium (3):
  - Research Site, Leuven
  - Research Site, Marchovelette
  - Research Site, Tessenderlo
- Brazil (8):
  - Research Site, Brasília
  - Research Site, Campinas
  - Research Site, Curitiba
  - Research Site, Fortaleza
  - Research Site, Joinville
  - Research SIte, Porto Alegre
  - Research Site, Recife
  - Research Site, São Paulo
- Canada (9):
  - Research Site, Coquitlam, British Columbia
  - Research Site, Penticton, British Columbia
  - Research Site, Ottawa, Ontario
  - Research Site, Gatineu, Quebec
  - Research Site, Mississauga
  - Research Site, Petitcodiac
  - Research Site, Pointe-Claire
  - Research Site, Regina
  - Research Site, Saint John
- France (4):
  - Research Site, Châteaugiron
  - Research Site, Mûrs-Erigné
  - Research Site, Nantes
  - Research Site, Vieux-Condé
- Germany (4):
  - Research Site, Dresden
  - Research Site, Mainz
  - Research Site, Münster
  - Research Site, Rodgau
- Hungary (4):
  - Research Site, Budapest
  - Research Site, Gyula
  - Research Site, Hódmezővásárhely
  - Research Site, Pécs
- India (7):
  - Research Site, Ahmedabad
  - Research Site, Bangalore
  - Research Site, Channai
  - Research Site, Kochi
  - Research Site, Mumbai
  - Research Site, New Dehli
  - Research SIte, Pune
- Israel (2):
  - Research Site, Holon
  - Research SIte, Tel Litwinsky
- Italy (3):
  - Research Site, Florence
  - Research Site, Milan
  - Research Site, Siena
- Mexico (3):
  - Research Site, Chihuahua City
  - Research Site, Guadalajara
  - Research Site, Monterrey
- Poland (3):
  - Research Site, Lublin
  - Research Site, Szczecin
  - Research Site, Wroclaw
- Puerto Rico (2):
  - Research Site, Manatí
  - Research Site, Toa Baja
- Romania (3):
  - Research Site, Galati
  - Research Site, Oradea
  - Research Site, Târgu Mureş
- Russia (5):
  - Research Site, Arkhangelsk
  - Research Site, Moscow
  - Research Site, Rostov-on-Don
  - Research Site, Saint Petersburg
  - Research Site, Stavropol
- Slovakia (2):
  - Research Site, Bratislava
  - Research Site, Trebišov
- South Africa (4):
  - Research Site, Johannesburg
  - Research Site, Kempton Park
  - Research Site, Midrand
  - Research Site, Soweto
- South Korea (5):
  - Research Site, Busan
  - Research Site, Daegu
  - Research Site, Jeonju
  - Research Site, Seoul
  - Research Site, Sungnam
- Spain (4):
  - Research Site, Alicante
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Seville
- Turkey (Türkiye) (3):
  - Research Site, Ankara
  - Research Site, Istanbul
  - Research Site, Sisli-Istanbul
- United Kingdom (8):
  - Research Site, Bath
  - Research Site, Birmingham
  - Research Site, Edinburgh
  - Research Site, Frome
  - Research Site, Guildford
  - Research Site, Hull
  - Research Site, Sheffield
  - Research Site, Swansea

REFERENCES:
- [Derived] Guja C, Frias JP, Suchower L, Hardy E, Marr G, Sjostrom CD, Jabbour SA. Safety and Efficacy of Exenatide Once Weekly in Participants with Type 2 Diabetes and Stage 2/3 Chronic Kidney Disease. Diabetes Ther. 2020 Jul;11(7):1467-1480. doi: 10.1007/s13300-020-00815-z. Epub 2020 Apr 18. PMID 32306296
- [Derived] Malloy J, Meloni A, Han J. Efficacy and tolerability of exenatide once weekly versus sitagliptin in patients with type 2 diabetes mellitus: a retrospective analysis of pooled clinical trial data. Postgrad Med. 2013 May;125(3):58-67. doi: 10.3810/pgm.2013.05.2661. PMID 23748507
- [Derived] Grimm M, Han J, Weaver C, Griffin P, Schulteis CT, Dong H, Malloy J. Efficacy, safety, and tolerability of exenatide once weekly in patients with type 2 diabetes mellitus: an integrated analysis of the DURATION trials. Postgrad Med. 2013 May;125(3):47-57. doi: 10.3810/pgm.2013.05.2660. PMID 23748506
- [Derived] Meloni AR, DeYoung MB, Han J, Best JH, Grimm M. Treatment of patients with type 2 diabetes with exenatide once weekly versus oral glucose-lowering medications or insulin glargine: achievement of glycemic and cardiovascular goals. Cardiovasc Diabetol. 2013 Mar 23;12:48. doi: 10.1186/1475-2840-12-48. PMID 23522121
- [Derived] Russell-Jones D, Cuddihy RM, Hanefeld M, Kumar A, Gonzalez JG, Chan M, Wolka AM, Boardman MK; DURATION-4 Study Group. Efficacy and safety of exenatide once weekly versus metformin, pioglitazone, and sitagliptin used as monotherapy in drug-naive patients with type 2 diabetes (DURATION-4): a 26-week double-blind study. Diabetes Care. 2012 Feb;35(2):252-8. doi: 10.2337/dc11-1107. Epub 2011 Dec 30. PMID 22210563

RESULTS

PARTICIPANT FLOW:
Groups:
- Exenatide Once Weekly: Exenatide once weekly (subcutaneous injection of 2 mg exenatide, once a week) + daily oral placebo
- Metformin: Metformin (1000 mg/day for 2 weeks, then 1500 mg/day for 2 weeks, then 2000 mg/day for 22 weeks) + weekly subcutaneous placebo injection
- Pioglitazone: Pioglitazone (30 mg/day for 4 weeks, then 45 mg/day for 22 weeks) + weekly subcutaneous placebo injection
- Sitagliptin: Sitagliptin (100 mg/day for 26 weeks) + weekly subcutaneous placebo injection
Period: Overall Study
Arm/Group | Exenatide Once Weekly | Metformin | Pioglitazone | Sitagliptin
Started | 248 | 246 | 163 | 163
Completed | 210 | 213 | 133 | 140
Not Completed | 38 | 33 | 30 | 23
Not completed — Adverse Event | 6 | 6 | 5 | 1
Not completed — Lost to Follow-up | 4 | 1 | 3 | 4
Not completed — Physician Decision | 3 | 3 | 2 | 3
Not completed — Protocol Violation | 5 | 9 | 2 | 5
Not completed — Withdrawal by Subject | 17 | 9 | 12 | 6
Not completed — Entry Criteria Not Met | 0 | 2 | 1 | 1
Not completed — Lack of Efficacy-Loss of Glucose Control | 3 | 3 | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exenatide Once Weekly | Metformin | Pioglitazone | Sitagliptin | Total
Number analyzed (Participants) | 248 | 246 | 163 | 163 | 820
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 217 | 215 | 135 | 144 | 711
  >=65 years | 31 | 31 | 28 | 19 | 109
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.7 (10.91) | 53.7 (11.08) | 55.3 (10.96) | 52.3 (11.05) | 53.7 (11.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109 | 92 | 66 | 69 | 336
  Male | 139 | 154 | 97 | 94 | 484
Glycosylated hemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of total hemoglobin] | 8.5 (1.19) | 8.6 (1.20) | 8.5 (1.24) | 8.5 (1.25) | 8.5 (1.22)
Weight [Mean (Standard Deviation); unit: kg] | 87.5 (18.88) | 85.9 (19.57) | 86.1 (17.77) | 88.7 (18.65) | 87.0 (18.83)

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c From Baseline to Week 26
Description: Change in HbA1c from baseline to Week 26.
Time Frame: Baseline, Week 26
Population: Intent to treat (ITT) population consisted of all randomized patients who had taken at least one dose of study drug. All scheduled post-baseline measurements were included in the analysis. Unscheduled visit observations were carried forward to the next scheduled visits.
Measure: Least Squares Mean (Standard Error); unit: percentage of total hemoglobin
Arm/Group | Exenatide Once Weekly | Metformin | Pioglitazone | Sitagliptin
Number analyzed (Participants) | 218 | 218 | 137 | 142
percentage of total hemoglobin | -1.53 (0.07) | -1.48 (0.07) | -1.63 (0.08) | -1.15 (0.08)
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Metformin; Power calculation: A sample of 740 (222 exenatide once weekly, 222 metformin, 148 pioglitazone, and 148 sitagliptin) would provide approximately 90% power to detect a true differences between exenatide once weekly and the 3 comparators: metformin, pioglitazone, and sitagliptin of 0.4%, 0.5%, and 0.5%, respectively in change in HbA1c from baseline to Week 26 with a 2-sided t test at a significance level of 0.05, assuming a common standard deviation of 1.2%; Test type: Non-Inferiority or Equivalence — Noninferiority Null Hypotheses: H1: The effect of exenatide is inferior to that of metformin. H2: The effect of exenatide is inferior to that of sitagliptin. H3: The effect of exenatide is inferior to that of pioglitazone. Then, the 3 superiority null hypotheses were tested. Change in HbA1c was analyzed using an MMRM analysis of covariance (ANCOVA) with treatment, baseline HbA1c, country, week of visit, and treatment-by week interaction as fixed effects; and patient and error as random effects; p = 0.620, Mixed Models Analysis — Noninferiority was tested by Bonferroni (margin 0.3%, adjusted significance of 0.0167). Superiority was tested by Hommel (nominal significance level was between 0.0167 and 0.05 depended on the number of noninferiority hypotheses rejected); Least Squares Mean Difference = -0.05, 98.3% CI 2-sided [-0.26 to 0.17], Standard Error of Mean 0.09
Statistical Analysis 2: Comparison: Exenatide Once Weekly vs Pioglitazone; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.328, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = 0.10, 98.3% CI 2-sided [-0.15 to 0.35], Standard Error of Mean 0.10
Statistical Analysis 3: Comparison: Exenatide Once Weekly vs Sitagliptin; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < .001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = -0.37, 98.3% CI 2-sided [-0.62 to -0.13], Standard Error of Mean 0.10

2. Primary Outcome: Percentage of Patients Achieving HbA1c <=7% at Week 26
Description: Percentage of patients achieving HbA1c <=7% at Week 26 (for patients with baseline HbA1c >7%).
Time Frame: Baseline, Week 26
Population: ITT subjects with baseline HbA1c>7%. Only patients with non-missing baseline value and at least one non-missing post-baseline value of the response variable were included in analysis. Missing data at endpoint was imputed using last observation carried forward (LOCF) approach.
Measure: Number; unit: percentage of patients
Arm/Group | Exenatide Once Weekly | Metformin | Pioglitazone | Sitagliptin
Number analyzed (Participants) | 226 | 232 | 150 | 143
percentage of patients | 64.2 | 57.3 | 63.3 | 45.5
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Metformin; Test type: Superiority or Other; p = 0.151, Fisher Exact — No multiple adjustment were done
Statistical Analysis 2: Comparison: Exenatide Once Weekly vs Pioglitazone; Test type: Superiority or Other; p = 0.913, Fisher Exact — No multiple adjustment were done
Statistical Analysis 3: Comparison: Exenatide Once Weekly vs Sitagliptin; Test type: Superiority or Other; p < .001, Fisher Exact — No multiple adjustment were done

3. Secondary Outcome: Change in Fasting Serum Glucose (FSG) From Baseline to Week 26
Description: Change in FSG from baseline to Week 26.
Time Frame: Baseline, Week 26
Population: ITT population. Only patients with non-missing baseline value and at least one non-missing post-baseline value of the response variable were included in analysis. All scheduled post-baseline measurements were included in the analysis, with no imputation of missing data other than that inherent in the MMRM model was used.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Exenatide Once Weekly | Metformin | Pioglitazone | Sitagliptin
Number analyzed (Participants) | 198 | 203 | 127 | 120
mmol/L | -2.25 (0.14) | -1.98 (0.14) | -2.57 (0.18) | -1.13 (0.18)
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Metformin; Change in FSG from baseline to Week 26 was analyzed using an MMRM ANCOVA model with treatment, baseline FSG, country, week of visit, and treatment-by week interaction as fixed effects; and patient and error as random effects; Test type: Superiority or Other; p = 0.155, Mixed Models Analysis — No multiple adjustment were done; Least Squares Mean Difference = -0.28, 95% CI 2-sided [-0.66 to 0.10], Standard Error of Mean 0.19
Statistical Analysis 2: Comparison: Exenatide Once Weekly vs Pioglitazone; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.153, Mixed Models Analysis — No multiple adjustment were done; Least Squares Mean Difference = 0.32, 95% CI 2-sided [-0.12 to 0.75], Standard Error of Mean 0.22
Statistical Analysis 3: Comparison: Exenatide Once Weekly vs Sitagliptin; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < .001, Mixed Models Analysis — No multiple adjustment were done; Least Squares Mean Difference = -1.12, 95% CI 2-sided [-1.56 to -0.68], Standard Error of Mean 0.22

4. Secondary Outcome: Change in Body Weight From Baseline to Week 26
Description: Change in Body Weight from baseline to Week 26.
Time Frame: Baseline, Week 26
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Exenatide Once Weekly | Metformin | Pioglitazone | Sitagliptin
Number analyzed (Participants) | 215 | 217 | 134 | 141
kg | -2.04 (0.21) | -2.00 (0.21) | 1.52 (0.26) | -0.76 (0.26)
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Metformin; Change in Body Weight from baseline to Week 26 was analyzed using an MMRM ANCOVA model with treatment, baseline body weight, country, week of visit, and treatment-by week interaction as fixed effects; and patient and error as random effects; Test type: Superiority or Other; p = 0.892, Mixed Models Analysis — No multiple adjustment were done; Least Squares Mean Difference = -0.04, 95% CI 2-sided [-0.61 to 0.53], Standard Error of Mean 0.29
Statistical Analysis 2: Comparison: Exenatide Once Weekly vs Pioglitazone; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < .001, Mixed Models Analysis — No multiple adjustment were done; Least Squares Mean Difference = -3.56, 95% CI 2-sided [-4.21 to -2.90], Standard Error of Mean 0.33
Statistical Analysis 3: Comparison: Exenatide Once Weekly vs Sitagliptin; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < .001, Mixed Models Analysis — No multiple adjustment were done; Least Squares Mean Difference = -1.28, 95% CI 2-sided [-1.92 to -0.63], Standard Error of Mean 0.33

5. Secondary Outcome: Change in Fasting Total Cholesterol (TC) From Baseline to Week 26
Description: Change in Fasting TC from baseline to Week 26.
Time Frame: Baseline, Week 26
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Exenatide Once Weekly | Metformin | Pioglitazone | Sitagliptin
Number analyzed (Participants) | 199 | 203 | 127 | 120
mmol/L | -0.24 (0.06) | -0.22 (0.06) | 0.09 (0.08) | -0.01 (0.08)
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Metformin; Change in Fasting TC from baseline to Week 26 was analyzed using an MMRM ANCOVA model with treatment, baseline TC, country, week of visit, and treatment-by week interaction as fixed effects; and patient and error as random effects; Test type: Superiority or Other; p = 0.873, Mixed Models Analysis — No multiple adjustment were done; Least Squares Mean Difference = -0.01, 95% CI 2-sided [-0.18 to 0.15], Standard Error of Mean 0.08
Statistical Analysis 2: Comparison: Exenatide Once Weekly vs Pioglitazone; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < .001, Mixed Models Analysis — No multiple adjustment were done; Least Squares Mean Difference = -0.33, 95% CI 2-sided [-0.52 to -0.14], Standard Error of Mean 0.10
Statistical Analysis 3: Comparison: Exenatide Once Weekly vs Sitagliptin; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.022, Mixed Models Analysis — No multiple adjustment were done; Least Squares Mean Difference = -0.22, 95% CI 2-sided [-0.41 to -0.03], Standard Error of Mean 0.10

6. Secondary Outcome: Change in Fasting High-Density Lipoprotein (HDL) From Baseline to Week 26
Description: Change in Fasting HDL from baseline to Week 26.
Time Frame: Baseline, Week 26
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Exenatide Once Weekly | Metformin | Pioglitazone | Sitagliptin
Number analyzed (Participants) | 199 | 203 | 127 | 120
mmol/L | 0.01 (0.01) | 0.07 (0.01) | 0.17 (0.02) | 0.04 (0.02)
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Metformin; Change in Fasting HDL from baseline to Week 26 was analyzed using an MMRM ANCOVA model with treatment, baseline HDL, country, week of visit, and treatment-by week interaction as fixed effects; and patient and error as random effects; Test type: Superiority or Other; p = 0.004, Mixed Models Analysis — No multiple adjustment were done; Least Squares Mean Difference = -0.05, 95% CI 2-sided [-0.09 to -0.02], Standard Error of Mean 0.02
Statistical Analysis 2: Comparison: Exenatide Once Weekly vs Pioglitazone; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p < .001, Mixed Models Analysis — No multiple adjustment were done; Least Squares Mean Difference = -0.15, 95% CI 2-sided [-0.19 to -0.11], Standard Error of Mean 0.02
Statistical Analysis 3: Comparison: Exenatide Once Weekly vs Sitagliptin; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.142, Mixed Models Analysis — No multiple adjustment were done; Least Squares Mean Difference = -0.03, 95% CI 2-sided [-0.07 to 0.01], Standard Error of Mean 0.02

7. Secondary Outcome: Ratio of Fasting Triglycerides at Week 26 to Baseline
Description: Ratio of Fasting Triglycerides (measured in mmol/L) at Week 26 to baseline. Log(Post-baseline Triglycerides) - log(Baseline Triglycerides); change from baseline to Week 26 is presented as ratio of endpoint to baseline.
Time Frame: Baseline, Week 26
Population: ITT population. Only patients with non-missing baseline value and at least one non-missing post-baseline value of the response variable were included in analysis. Missing data at endpoint was imputed using LOCF approach.
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Exenatide Once Weekly | Metformin | Pioglitazone | Sitagliptin
Number analyzed (Participants) | 200 | 204 | 127 | 121
ratio | 0.98 (0.03) | 0.96 (0.03) | 0.85 (0.03) | 0.94 (0.04)
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Metformin; Fasting triglycerides data were logarithm-transformed and the change at Week 26 to baseline, expressed as the ratio, was analyzed using ANCOVA model with treatment and country as factors and baseline triglycerides as a covariate; Test type: Superiority or Other; p = 0.657, ANCOVA — No multiple adjustment were done; Geometric Least Squares Mean Ratio = 1.02, 95% CI 2-sided [0.94 to 1.10], Standard Error of Mean 0.04
Statistical Analysis 2: Comparison: Exenatide Once Weekly vs Pioglitazone; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.002, ANCOVA — No multiple adjustment were done; Geometric Least Squares Mean Ratio = 1.16, 95% CI 2-sided [1.06 to 1.27], Standard Error of Mean 0.05
Statistical Analysis 3: Comparison: Exenatide Once Weekly vs Sitagliptin; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.398, ANCOVA — No multiple adjustment were done; Geometric Least Squares Mean Ratio = 1.04, 95% CI 2-sided [0.95 to 1.14], Standard Error of Mean 0.05

8. Secondary Outcome: Assessment on Event Rate of Treatment-emergent Major Hypoglycemic Events
Description: Major hypoglycemia is defined as any event that has symptoms consistent with hypoglycemia resulting in loss of consciousness or seizure that shows prompt recovery in response to administration of glucagon or glucose, or documented hypoglycemia (blood glucose <3.0 mmol/L [54 mg/dL]) requiring the assistance of another person because of severe impairment in consciousness or behavior (whether or not symptoms of hypoglycemia are detected by the patient). Mean event rate = total number of events for all subjects in a treatment regimen / the total number of subject years of exposure for all subjects in that treatment. Standard error = square root of (total number of events / (subject years of exposure)**2).
Time Frame: Baseline to Week 26
Population: ITT population.
Measure: Mean (Standard Error); unit: events per subject-year
Arm/Group | Exenatide Once Weekly | Metformin | Pioglitazone | Sitagliptin
Number analyzed (Participants) | 248 | 246 | 163 | 163
events per subject-year | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000)

9. Secondary Outcome: Assessment on Event Rate of Treatment-Emergent Minor Hypoglycemic Events
Description: Minor hypoglycemia is defined as a sign or symptom associated with hypoglycemia that is either self-treated by the patient or resolves on its own AND has a concurrent finger stick blood glucose <3.0 mmol/L (54 mg/dL) and not classified as major hypoglycemia. Mean event rate = total number of events for all subjects in a treatment regimen / the total number of subject years of exposure for all subjects in that treatment. Standard error = square root of (total number of events / (subject years of exposure)**2).
Time Frame: Baseline to Week 26
Population: ITT population.
Measure: Mean (Standard Error); unit: events per subject-year
Arm/Group | Exenatide Once Weekly | Metformin | Pioglitazone | Sitagliptin
Number analyzed (Participants) | 248 | 246 | 163 | 163
events per subject-year | 0.05 (0.021) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000)

10. Secondary Outcome: Change in Systolic Blood Pressure From Baseline to Week 26.
Description: Change in Systolic Blood Pressure from baseline to Week 26.
Time Frame: Baseline, Week 26
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Exenatide Once Weekly | Metformin | Pioglitazone | Sitagliptin
Number analyzed (Participants) | 215 | 217 | 134 | 141
mmHg | -1.25 (0.79) | 0.14 (0.78) | -1.74 (0.98) | -1.81 (0.96)
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Metformin; Change in Systolic Blood Pressure from baseline to Week 26 was analyzed using an MMRM ANCOVA model with treatment, baseline systolic blood pressure, country, week of visit, and treatment-by week interaction as fixed effects; and patient and error as random effects; Test type: Superiority or Other; p = 0.201, Mixed Models Analysis — No multiple adjustment were done; Least Squares Mean Difference = -1.39, 95% CI 2-sided [-3.52 to 0.74], Standard Error of Mean 1.09
Statistical Analysis 2: Comparison: Exenatide Once Weekly vs Pioglitazone; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p = 0.693, Mixed Models Analysis — No multiple adjustment were done; Least Squares Mean Difference = 0.49, 95% CI 2-sided [-1.94 to 2.93], Standard Error of Mean 1.24
Statistical Analysis 3: Comparison: Exenatide Once Weekly vs Sitagliptin; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p = 0.646, Mixed Models Analysis — No multiple adjustment were done; Least Squares Mean Difference = 0.56, 95% CI 2-sided [-1.84 to 2.96], Standard Error of Mean 1.22

11. Secondary Outcome: Change in Diastolic Blood Pressure From Baseline to Week 26.
Description: Change in Diastolic Blood Pressure from baseline to Week 26.
Time Frame: Baseline, Week 26
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Exenatide Once Weekly | Metformin | Pioglitazone | Sitagliptin
Number analyzed (Participants) | 215 | 217 | 134 | 141
mmHg | -0.50 (0.51) | -0.86 (0.50) | -2.50 (0.63) | -0.45 (0.62)
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Metformin; Change in Diastolic Blood Pressure from baseline to Week 26 was analyzed using an MMRM ANCOVA model with treatment, baseline diastolic blood pressure, country, week of visit, and treatment-by week interaction as fixed effects; and patient and error as random effects; Test type: Superiority or Other; p = 0.610, Mixed Models Analysis — No multiple adjustment were done; Least Squares Mean Difference = 0.36, 95% CI 2-sided [-1.02 to 1.73], Standard Error of Mean 0.70
Statistical Analysis 2: Comparison: Exenatide Once Weekly vs Pioglitazone; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.013, Mixed Models Analysis — No multiple adjustment were done; Least Squares Mean Difference = 2.00, 95% CI 2-sided [0.43 to 3.58], Standard Error of Mean 0.80
Statistical Analysis 3: Comparison: Exenatide Once Weekly vs Sitagliptin; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.946, Mixed Models Analysis — No multiple adjustment were done; Least Squares Mean Difference = -0.05, 95% CI 2-sided [-1.60 to 1.49], Standard Error of Mean 0.79

ADVERSE EVENTS:
Arm/Group | Exenatide Once Weekly | Metformin | Pioglitazone | Sitagliptin
Serious Adverse Events (participants affected / at risk) | 4/248 | 12/246 | 9/163 | 3/163
Other Adverse Events (participants affected / at risk) | 109/248 | 94/246 | 57/163 | 55/163
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Exenatide Once Weekly (N=248) | Metformin (N=246) | Pioglitazone (N=163) | Sitagliptin (N=163)
Calculus ureteric (Renal and urinary disorders) | 1 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Joint sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 1 | 0 | 0
Arteriovenous malformation (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Arteritis (Vascular disorders) | 0 | 0 | 0 | 1
Arthritis bacterial (Infections and infestations) | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0
Chondromalacia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Diabetic foot (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Hysterectomy (Surgical and medical procedures) | 0 | 1 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1 | 0 | 0
Lumbar hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Oedema (General disorders) | 0 | 0 | 1 | 0
Peritonsillar abscess (Infections and infestations) | 0 | 1 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Typhoid fever (Infections and infestations) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Wound infection (Infections and infestations) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Exenatide Once Weekly (N=248) | Metformin (N=246) | Pioglitazone (N=163) | Sitagliptin (N=163)
Nausea (Gastrointestinal disorders) | 28 | 17 | 6 | 6
Diarrhoea (Gastrointestinal disorders) | 27 | 31 | 6 | 9
Injection site nodule (General disorders) | 26 | 25 | 6 | 11
Constipation (Gastrointestinal disorders) | 21 | 8 | 3 | 4
Headache (Nervous system disorders) | 20 | 30 | 13 | 15
Nasopharyngitis (Infections and infestations) | 19 | 11 | 14 | 16
Dyspepsia (Gastrointestinal disorders) | 18 | 8 | 8 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 | 3 | 5 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 14 | 7 | 5
Hypertension (Vascular disorders) | 3 | 3 | 12 | 3
Oedema peripheral (General disorders) | 0 | 1 | 12 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days